CLINICAL TRIAL: NCT07175714
Title: Evaluating Methods to Replicate Stumbles and Slips During Walking
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Collaborators: University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CIP2024100353
Record Dates: First submitted 2025-08-06; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Fall Prevention; Balance, Falls; Amputation of Lower Limb
Keywords: amputation; falls; fall prevention; balance

STUDY DESIGN:
Masking Description: Able-Bodied Individuals Arm Prosthetic Users Arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Able-Bodied Individuals Arm (Experimental): Able-bodied subjects will undergo the same series of gait perturbation tests for comparison of adaptive gait responses.
  Interventions: Other: Methodologies to induce gait perturbations
- Prosthetic Users (Experimental): Amputee subjects will undergo a series of gait perturbation tests to evaluate adaptive responses.
  Interventions: Other: Methodologies to induce gait perturbations

INTERVENTIONS:
Other: Methodologies to induce gait perturbations — Method 1: Obstacles deployed at the frond end side of the treadmill Method 2: Obstacles deployed on the side of the treadmill Method 3: Spit-bell treadmill to induce slip perturbations Method 4: String method

SUMMARY:
This protocol outlines a study designed to investigate three different methodologies for inducing gait perturbations.

Subjects will be divided into two groups: prosthetic users and able-bodied individuals.

Each group will undergo a series of tests where controlled perturbations are applied using up to three methodologies with the number depending on factors such as time and fatigue. These methodologies may include mechanical, visual, or auditory perturbations designed to mimic unexpected obstacles or changes in terrain.

ELIGIBILITY:
Inclusion Criteria:

* 40 kg < body weight < 136kg
* Cognitive ability to understand all instructions and questionnaires in the study
* Willing and able to participate in the study and following the protocol
* Age ≥ 18 years
* Able to walk independently without the use of assistive device such as a cane or walker
* Able-bodied subjects OR Regular prosthesis users for at least 1 year with unilateral lower limb amputation at or below the transfemoral level (or equivalent level limb deficiency)

Exclusion Criteria:

* Subjects with pain which can affect their mobility
* Users with socket comfort score less than 7
* Subjects with cognitive impairment
* Pregnant subjects
* Musculoskeletal disorders or neurological conditions that affect motor function, gait or balance
* Use of medications that are known to impair balance and coordination
* Any other conditions deemed by the investigator to make participation unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Gait Perturbation Methods in Inducing Stumble or Fall Events | For each gait perturbation method, events are assessed during its application within a single testing session (approximately 30-60 minutes); multiple methods may be tested per session.
  This measure evaluates the effectiveness of various gait perturbation methodologies in successfully inducing perturbation events that result in stumbles or falls. Data will be collected on the number of perturbation events, with a particular focus on those leading to stumbles or falls. The incidence rate will be calculated as the number of perturbation events resulting in stumbles or falls per total number of perturbations. The target outcome is for at least 80% of perturbations to create an event that results in a stumble or fall. Descriptive statistics will be used to summarize the findings and assess the overall effectiveness of the perturbation methods.
Subjective Evaluation of Gait Perturbation Methodologies | Participant feedback is collected immediately after each gait perturbation method within a single testing session (approximately 30-60 minutes); multiple methods may be evaluated per session.
  This measure focuses on assessing participant feedback regarding the effectiveness and realism of different gait perturbation methodologies. Participants will provide ratings based on a questionnaire, excluding safety-related questions, to capture their experiences and perceptions. The goal is for all subjects to rate the methodologies as at least neutral or safe. Descriptive statistics will be employed to analyze the ratings, offering valuable insights into user experiences and perceptions of the perturbation methods.
Safety Perception of Gait Perturbation Methodologies | Participant feedback is collected immediately after each gait perturbation method within a single testing session (approximately 30-60 minutes); multiple methods may be evaluated per session.
  This measure evaluates participants' perceptions of safety regarding the gait perturbation methodologies used in the study. Participants will provide ratings based on a specific safety question from a questionnaire. The aim is for all subjects to rate the safety of the methods as at least neutral or safe. Descriptive statistics will be used to summarize the feedback, ensuring that the perturbation methods are perceived as minimizing the risk of injury and maintaining participant safety.
Unpredictability of Gait Perturbation Methodologies | Participant feedback is collected immediately after each gait perturbation method within a single testing session (approximately 30-60 minutes); multiple methods may be evaluated per session.
  This measure assesses the extent to which gait perturbation events are unnoticed and unexpected by participants. Feedback will be collected after each perturbation event, using a yes/no question to determine whether participants anticipated the perturbation. The objective is for at least 90% of perturbations to be perceived as unnoticed and unexpected. Descriptive statistics will be utilized to analyze the data, providing insights into the effectiveness of the methodologies in creating genuinely unpredictable perturbation events.
Consistency of Gait Perturbation Incidence Rates Over Time | For each gait perturbation method, events are assessed during its application within a single testing session (approximately 30-60 minutes); multiple methods may be tested per session.
  This measure evaluates the consistency of incidence rates for perturbation events among able-bodied subjects over time. The focus is on comparing the incidence rates of stumbles or falls from the first two perturbations to the last two perturbations. The goal is to ensure that the methodologies lead to a similar number of incidents throughout the study, with no more than a 10% difference observed between these two sets of perturbations. Descriptive statistics will be used to assess the data, ensuring stability and reliability in the perturbation methodologies across the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Thor Fridriksson, Doctor, Principal Investigator — Össur Iceland ehf
Locations (2):
- Iceland (2):
  - University of Iceland, Reykjavik
  - Össur Iceland ehf., Reykjavik

IPD SHARING:
Plan to Share IPD: No